CLINICAL TRIAL: NCT06477146
Title: Pilot Study of Milk Thistle for the Treatment of Pediatric Non-Alcoholic Fatty Liver Disease (NAFLD)
Brief Title: Milk Thistle Clinical Trial in Pediatric NAFLD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Thomas J Sferra, MD, Pediatric Gastroenterology, Division Chief, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY20231215
Record Dates: First submitted 2024-06-20; First posted 2024-06-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Non-Alcoholic Fatty Liver Disease (NAFLD)
Keywords: Silymarin; Fatty Liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver | interventions — milk-thistle extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Milk Thistle (Experimental): Patients will be given Milk Thistle capsules based on weight by mouth once or twice daily for 12 weeks.
  Interventions: Drug: Milk thistle (MT); Behavioral: Lifestyle Modification; Device: Fibroscan
- Placebo (Experimental): Patients will be give 500mg capsule based on weight by mouth once or twice daily for 12 weeks.
  Interventions: Drug: Placebo; Behavioral: Lifestyle Modification; Device: Fibroscan

INTERVENTIONS:
Drug: Milk thistle (MT) — MT capsules will contain 300 mg of MT with 80% content of Silymarin, standardized to 240mg Silymarin content. Dosing will be based on body weight with maximum dose of 600 mg/day. Dosing will be either 1 or 2 capsules per day based on weight.
  Arms: Milk Thistle
Drug: Placebo — The placebo is consistent of Psyllium husk fiber, in 500mg per capsule composition.
  Arms: Placebo
Behavioral: Lifestyle Modification — The primary instructions for lifestyle modification are:
  1. Physical activity goal- 20-30 minutes per day 5 to 7 days per week. The aim is 150 minutes a week and more than 300 calories burnt for each workout.
  2. Adequate hydration- 4-5 bottles of water a day.
  3. Limitation of sugar-free beverages- once daily and 1-2 (8 oz) cups of skim/1% milk (or dairy alternative) daily.
  4. Avoidance of beverages with added sugar such as soda, Kool-Aid, juice, and Gatorade.
  5. Ideal consumption- three meals daily(breakfast, lunch, dinner)and one snack.
  6. Snack Goal <200 calories. If a 2nd, 3rd, etc. snack is desired it will only be a vegetable.
  7. Five servings of fruits/vegetables per day.
  8. Each food we recommend eating should have dietary fiber >3 grams/serving. Ideally >5 grams/serving.
  9. The given survival guide will have all information regarding serving size and portion allotment.
  10. "MyPlate.gov" handout given which will guide participants in relation to portion control.
Device: Fibroscan — FibroScan will be completed to measure Elastography. Elastography works by emitting small pulse of energy which may be perceived as a vibration which quickly calculated the stiffness of the liver, which correlates to fat deposition and fibrosis.

SUMMARY:
Pediatric Fatty Liver disease is a growing problem in the United States and is expected to be the leading cause of Liver Transplantation in Adults in 20 years. Following lifestyle changes such as diet restrictions and exercise may be difficult to consistently maintain. The purpose of this study is to investigate alternative medical therapy with an herbal supplement called Milk Thistle (MT) which may improve fatty liver disease and would be easier to follow than diet and exercise.

ELIGIBILITY:
Inclusion Criteria:

Subjects between the age of 9 to 22 years old diagnosed with non-Alcoholic Fatty Liver Disease (NAFLD) based on current North American Society for Pediatric Gastroenterology, Hepatology and Nutrition Guidelines:

* a. Elevated ALT levels greater than 2 times the sex specific upper limit of normal at baseline; (for boys ALT greater than 50 U/L, and girls ALT greater than 44 U/L) i. AND either overweight (with risk factors as noted below) or obese children:

  * 1. In children, obesity is defined as BMI greater than or equal to 95th percentile in weight and overweight is defined as greater than or equal to the 85th percentile to less than the 95th percentile.
  * 2. Risk factors associated with overweight child that warrant screening and inclusion are:

    a. Central obesity, Family history of NAFLD/non-alcoholic steatohepatitis(NASH), pre-diabetic or diabetic, dyslipidemia, sleep apnea)
  * 3. For participants 18 years or older: Obesity is defined as BMI greater than or equal to 30 kg/m2; overweight is defined as BMI greater than or equal to 25 kg/m2 and less than 30 kg/m2.
* b. Evidence of Sonographic presence of hepatic steatosis with greater than 5% steatosis on Ultrasound or FibroScan [with a controlled attenuation parameter (CAP) score of 238 or greater)] prior to start of trial starting.
* c. (Or) previous findings on Liver Biopsy consistent with NAFLD including hepatic macro-vesicular steatosis, ballooning degeneration or Mallory Denk Bodies

Contraception Requirements for Enrollment of adult population:

1. Female participants are eligible if the participant is of reproductive potential and have a negative -serum pregnancy test (beta human chorionic gonadotropin), are not breastfeeding, and do not plan to become pregnant during the study and agree to use two highly effective birth control methods during the study OR if the participant is not of child-bearing potential (i.e., surgically [bilateral oophorectomy, hysterectomy, or tubal ligation] or naturally sterile [> 12 consecutive months without menses]).

   Highly effective birth control methods include condoms with spermicide, diaphragm with spermicide, hormonal and nonhormonal intrauterine device, hormonal contraception (estrogens stable ≥ 3 months), a vasectomized male partner, or sexual abstinence (defined as refraining from heterosexual intercourse), from screening, throughout the study, and for at least 30 days after the last dose of study drug administration. Reliance on abstinence from heterosexual intercourse is acceptable only if it is the patient's habitual practice.
2. Male patients who are sexually active with a partner of child-bearing potential must either be sterile (vasectomy with history of a negative sperm count at least 90 days following the procedure); practice total abstinence from sexual intercourse as the preferred lifestyle (periodic abstinence is not acceptable); use a male condom with any sexual activity; or agree to use a birth control method considered to be appropriate by the Investigator (such as one of the methods identified above for female patients of childbearing potential) from the time of screening until 30 days after the last dose of study drug administration. Male patients must agree not to donate sperm for a period of 30 days after the last dose of study drug administration.

Exclusion Criteria:

1. Patients with cardiovascular disorders (such as history of myocardial infarction, stroke, DVT)
2. Medical conditions including history of malignancy, transplantation, immunologic diseases (rheumatoid arthritis, inflammatory bowel disease, systemic lupus erythematosus, autoimmune thyroiditis, idiopathic thrombocytopenic purpura, autoimmune hemolytic anemia, severe psoriasis, rheumatoid arthritis etc.), poorly controlled thyroid disease, uncontrolled hypertension.
3. Patients with cirrhosis and hepatic decompensation will be excluded from the study. Hepatic biomarker parameters will be excluded:

   * ALT greater than 200 U/L
   * AST greater than 200 U/L
   * Total bilirubin greater than 2.0 mg/dL
   * ALP greater than 500 U/L
   * INR greater than 1.4
   * GGT greater than 200 U/L
4. Subjects with history or other evidence of severe illness or any other conditions that would make the subject, in the opinion of the investigator, unsuitable for participation in the trial (such as poorly controlled psychiatric illness).
5. Subjects with unstable diabetes, or HbA1c >9% will be excluded from the study.
6. Subjects who report binge drinking will be excluded from this study.
7. Subjects who partake or state consumption history of tobacco use, vaping, marijuana use, or illicit drug abuse will be excluded from the study.
8. Subjects with severe hepatic dysfunction and synthetic dysfunction with hypoalbuminemia (Albumin < 3.0 g/dL), thrombocytopenia (platelet count <140,000/ml3), or coagulopathy (INR >1.4) will be excluded from the study.
9. Exclude subjects with abnormal renal function characterized as serum creatinine greater than the upper limit of normal range (based on the University of Iowa, Department of Pathology Lab Services Handbook):

   Pediatric Age Group Premature 0.3 - 1.0 mg/dL Neonates 0.2 - 0.9 mg/dL 2-12 months 0.2 - 0.4 mg/dL 1-2 years 0.2 - 0.5 mg/dL 3-4 years 0.3 - 0.7 mg/dL 5-6 years 0.3 - 0.7 mg/dL 7-8 years 0.2 - 0.6 mg/dL 9-10 years 0.3 - 0.7 mg/dL 11-12 years 0.3 - 0.9 mg/dL 13-15 years 0.4 - 0.9 mg/dL

   Males 16 years and older 0.6 - 1.2 mg/dL Females 16 years and older 0.5 - 1.0 mg/dL
10. Breast feeding women will be excluded from this clinical trial.
11. Subjects who are participating in other drug trials will be excluded from participating.
12. Subjects with a reported or known history of allergy or anaphylactic reaction to Ragweed will be excluded from this study.

Ages: 9 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Hepatic biomarker alanine aminotransferase (ALT) as measured by blood test. | Up to 12 weeks
Hepatic Stiffness (kilopascal, kPa) as measured by FibroScan. | Up to 12 weeks
  Normal kPa results are usually between 2 and 7 kPa, with the highest possible result of 75 kPa.
Percent of Hepatic Steatosis as measured by FibroScan. | Up to 12 weeks
  Percentage of steatosis will be correlated with the CAP score- 200 to 400db/m2

SECONDARY OUTCOMES:
Number of adverse events as measured by patient report. | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Sferra, MD, Principal Investigator — University Hospitals
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No